CLINICAL TRIAL: NCT04366154
Title: Impact of the COVID-19 Infectious Epidemic on the Management of Oncology and Onco-hematology Patients and on the Psychological Consequences for Patients and Caregivers
Acronym: COVIPACT
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-A00879-30
Record Dates: First submitted 2020-04-16; First posted 2020-04-28 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: COVID-19; Cancer
MeSH Terms: conditions — COVID-19; Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients
  Interventions: Other: Questionnaire
- Caregivers
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — delivery of questionnaires on perceived stress, post-traumatic stress, sleep disorders, quality of life, cognitive complaint

SUMMARY:
This original study will assess the impact of the coronavirus health crisis on the management of patients undergoing medical treatment for cancer, in particularly on the modification of the hospital organization. It will also provide a record of the progress of patients who will have been treated during the epidemic period and infected by the virus.

We will also assess the psychological impact of the pandemic in patients but also in caregivers

ELIGIBILITY:
Inclusion Criteria:

For Patients:

* Adult patient, treated for a solid or hematological tumor
* will be treated ou actually treated by oncological treatment carried out at the hospital in day unit of the participating centers: treatment initiated before or during the pandemic with COVID-19

For the Caregivers:

- Medical oncologist, hematologist, intern, nurse and caregiver in day unit of hospital

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 2 populations were recruted in this study : patients with cancer and caregivers
Sampling Method: Probability Sample
Enrollment: 809 (Actual)
Dates: Start 2020-04-15 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
To assess the impact of the COVID-19 pandemic on the modifications of treatments administered in hospital (day units) to patients with cancer or malignant hemopathy | up to 6 months
  Proportion of patients with modification of the treatments administered
To assess the impact of the COVID-19 pandemic on the change in the rate of treatment administration in hospital (day units) to patients with cancer or malignant hemopathy | up to 6 months
  Proportion of patients with change in the rate of treatment administration
To assess the impact of the COVID-19 pandemic on the number of cures administeredin hospital (day units) to patients with cancer or malignant hemopathy | up to 6 months
  Proportion of patients with change in the number of cures administered
To assess the impact of the COVID-19 pandemic on change of modality of administration in hospital (day units) to patients with cancer or malignant hemopathy | up to 6 months
  Proportion of patients with change of modality of administration (home administration to replace day hospital administration, teleconsultation uses)

SECONDARY OUTCOMES:
Evaluate the perceived stress on cancer patients treated in unit day of hospital | up to 12 months
  Score of questionnaires of Perceived Stress Scale [0-40 points]
Evaluate the post-traumatic stress on cancer patients treated in unit day of hospital | up to 12 months
  Score of questionnaires of Impact of Event Scale-Revised [0-88 points]
Evaluate the sleep disorders on cancer patients treated in unit day of hospital | up to 12 months
  Score of questionnaires of sleep disorders (ISI scale, 0-28 points)
Evaluate the quality of life on cancer patients treated in unit day of hospital | up to 12 months
  Score of questionnaires of quality of life (FACT-G scale)
Evaluate the cognitive complaints on cancer patients treated in unit day of hospital | up to 12 months
  Score of questionnaires of cognitive complaints (Fact-Cog scales; 0-148 points)
Evaluate the perceived stress on caregivers (perceived stress, post-traumatic stress, burnout, feeling of personal effectiveness) | up to 12 months
  Score of questionnaires of Perceived Stress Scale [0-40 points]
Evaluate the post-traumatic stress on caregivers (perceived stress, post-traumatic stress, burnout, feeling of personal effectiveness) | up to 12 months
  Score of questionnaires of Impact of Event Scale-Revised [0-88 points]
Evaluate the burnout on caregivers (perceived stress, post-traumatic stress, burnout, feeling of personal effectiveness) | up to 12 months
  Score of questionnaires of burnout ((Maslach Burn Out Inventory scale, 0-132 points)
Evaluate the feeling of personal effectiveness on caregivers (perceived stress, post-traumatic stress, burnout, feeling of personal effectiveness) | up to 12 months
  Score of questionnaires of feeling of personal effectiveness (0-30 points)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Centre François Baclesse, Caen
  - Centre Henri Becquerel, Rouen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cherifi F, Gernier F, Jardin F, Lefevre-Arbogast S, Bastien E, Lequesne J, Rigal O, Quilan F, Clarisse B, Grellard JM, Binarelli G, Fernette M, Lange M, Richard D, Morel A, Griffon B, Pepin LF, Leconte A, Faveyrial A, Leheurteur M, Beauplet B, Joly F. Post-traumatic stress disorder symptoms and quality of life among older patients with cancer during the COVID-19 pandemic. J Geriatr Oncol. 2023 Nov;14(8):101634. doi: 10.1016/j.jgo.2023.101634. Epub 2023 Sep 25. PMID 37757587
- [Derived] Bastien E, Lefevre-Arbogast S, Lequesne J, Gernier F, Cherifi F, Rigal O, Guittet L, Grellard JM, Binarelli G, Lange M, Fernette M, Tron L, Morel A, Richard D, Griffon B, Leconte A, Quilan F, Pepin LF, Jardin F, Leheurteur M, Faveyrial A, Clarisse B, Joly F. Posttraumatic Stress Symptoms in Patients With Cancer During the COVID-19 Pandemic: A One-Year Longitudinal Study. J Natl Compr Canc Netw. 2023 Feb 22;21(3):265-272.e7. doi: 10.6004/jnccn.2023.7085. PMID 36812938